CLINICAL TRIAL: NCT07005427
Title: Development of Dysphagia Management Protocol for Adult Patients in Intensive Care Unit
Brief Title: Comparison of Traditional Dysphagia Therapy and Developed Protocol for Dysphagia Patients in Intensive Care Unit
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Anum Ashraf REC/RCR & AHS/22
Record Dates: First submitted 2025-05-15; First posted 2025-06-05 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Dysphagia
Keywords: Dysphagia; ICU; Management Protocol
MeSH Terms: conditions — Deglutition Disorders | interventions — Guidelines as Topic

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Comparison group (Active Comparator): This Group will receive traditional dysphagia therapy.
  Interventions: Other: dysphagia therapy
- Experimental Group (Experimental): This group will receive treatment as per recently designed dysphagia management protocol, that includes the role of early mobilization, dietary intervention with varying postures, and overall care designed for first 48 hours.
  Interventions: Behavioral: Designed protocol for dysphagia

INTERVENTIONS:
Other: dysphagia therapy — This group will receive usual dysphagia care as provided in ICU settings
  * Standard bedside swallowing evaluation
  * Conventional compensatory strategies (postural changes, diet modifications)
  * Traditional exercises focusing on oral motor control
  * Therapy sessions 3 times per week for 30 minutes
  Other Names: traditional dysphagia therapy
  Arms: Comparison group
Behavioral: Designed protocol for dysphagia — * Innovative strengthening exercises adapted for ICU setting
  * Early mobilization component
  * ICU-specific compensatory strategies
  * Therapy sessions 5 times per week for 30 minutes with additional brief daily reinforcement
  Other Names: Guidelines
  Arms: Experimental Group

SUMMARY:
Dysphagia (swallowing disorders) in intensive care unit (ICU) patients is associated with poor outcomes, including aspiration pneumonia, prolonged hospitalization, and increased mortality. Traditional dysphagia management approaches may be insufficient for the unique needs of critically ill patients. This study aims to evaluate the effectiveness of a newly developed ICU-specific dysphagia protocol compared to traditional therapy approaches.

DETAILED DESCRIPTION:
The aim of this study are:

1. To compare the efficacy of traditional dysphagia therapy versus a developed ICU-specific protocol in improving swallowing function
2. To assess the impact of both approaches on clinical outcomes including aspiration rates, time to oral intake, ICU length of stay, and pneumonia incidence
3. To identify patient subgroups that may benefit most from the specialized protocol Methods Study Design

   * Prospective randomized controlled trial
   * Single-center study in a tertiary hospital ICU
   * 1:1 randomization to intervention or control group Participants
   * Total sample size: 90 adult ICU patients (45 per group)
   * Inclusion criteria: Adult patients (≥18 years) admitted to ICU with confirmed dysphagia by bedside evaluation within 72 hours of admission
   * Exclusion criteria: Preexisting neurological disorders affecting swallowing, head and neck cancer, inability to follow commands, expected ICU stay <48 hours This study will provide evidence for the efficacy of a specialized dysphagia management protocol tailored to the unique needs of critically ill patients. If proven effective, the protocol could establish new standards of care for dysphagia management in ICU settings, potentially improving patient outcomes and reducing healthcare costs associated with dysphagia-related complications.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (≥18 years) admitted to ICU with confirmed dysphagia by bedside evaluation within 72 hours of admission
* GCS more then 8

Exclusion Criteria:

* Preexisting neurological disorders affecting swallowing, head and neck cancer, inability to follow commands, expected ICU stay <48 hours

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2025-07-02 (Actual); Primary Completion 2026-04-16 (Estimated); Study Completion 2026-05-10 (Estimated)

PRIMARY OUTCOMES:
Improved Swallow Capacity | 6 months
  • Change in Functional Oral Intake Scale (FOIS) score from baseline to discharge (at discharge it should be more then 5 on its rating scale)

SECONDARY OUTCOMES:
Improved Quality of Life | 4 months
  • Patient satisfaction with swallowing function

CONTACTS AND LOCATIONS:
Overall Officials: Anum Ashraf, PhD*, Principal Investigator — Riphah International University; Nazia Mumtaz, PhD*, Study Director — Riphah International University
Locations (1):
- Riphah International University Lahore Campus, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No